CLINICAL TRIAL: NCT06971133
Title: Causes of Secondary and Prolonged Fever During Treatment of Bacterial Meningitis and Viral Encephalitis
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Kerolos Atef Shafeek Tanious, Doctor, Assiut University
Other Study IDs: meningitis and encephalitis
Record Dates: First submitted 2025-04-29; First posted 2025-05-14 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Meningitis in Children; Encephalitis in Children

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the present study is to investigate causes of secondary and prolonged fever during treatment of viral encephalitis and bacterial meningitis in children aged from one month to 18 years .

DETAILED DESCRIPTION:
Fever is a common symptom in both viral encephalitis and bacterial meningitis. However, in some patients, fever may persist or recure during the course of treatment. This can be concerning and may indicate unresolved infection, secondary infections, inflammatory responses, or treatment complications. Understanding the underlying causes and adopting a structured approach to management is crucial for improving patient care. Prolonged fever means fever persisting beyond 8-10 days despite appropriate treatment. Secondary fever means fever occurring after an initial period of defervescence, meaning the fever had initially subsided for at least 48 hours before recurring or a new fever spike following an apparent resolution. The common and established causes of secondary and prolonged fever in pediatrics patients during the treatment of bacterial meningitis and viral encephalitis include, nosocomial infections, subdural effusion, phlebitis, pneumonia , drug fever, otitis media, gastroenteritis and urinary tract infection . Subdural effusion prolongs fever in patients with meningitis. It occurs as a complication due to persistent inflammation, secondary infection, or inadequate resolution of the infection within the subdural space. Urinary tract infections (especially in catheterized patients) is nosocomial or superimposed infections that cause secondary or prolonged fever in pediatric patients during the treatment of meningitis or encephalitis. Otitis media can cause secondary or prolonged fever during the treatment of meningitis and encephalitis in pediatric patients. This can occur due to persistent infection, suppurative complications (such as mastoiditis or subdural empyema), or an inadequate response to initial antimicrobial therapy. Pneumonia, including hospital-acquired pneumonia, can cause secondary or prolonged fever during the treatment of CNS infections in pediatric patients. This occurs due to superimposed bacterial infections, ventilator-associated pneumonia in critically ill children, or aspiration pneumonia in patients with neurological compromise. Gastro-entritis can occur in hospitalized children undergoing treatment for CNS infections due to concurrent infections, dehydration-related metabolic disturbances, or systemic inflammatory responses. Enteric pathogens such asRotavirus, Norovirus, or bacterial causes like Salmonella and Clostridioides difficile can contribute to prolonged fever in hospitalized children undergoing treatment for CNS infections. Phlebitis can cause secondary fever during the treatment of encephalitis and meningitis in pediatric patients. It is often associated with intravenous catheter use, leading to localized or systemic infections, including catheterrelated bloodstream infections, which can contribute to persistent or recurrent fever.

Drug fever is a well-recognized phenomenon where fever arises as an adverse reaction to medications, often without an identifiable infectious source. It typically resolves upon discontinuation of the offending drug. In the context of meningitis and encephalitis treatment, antibiotics (e.g., beta-lactams, sulfonamides, vancomycin), anticonvulsants, and antipyretics have been implicated. A relapse of encephalitis or meningitis occurs due to incomplete eradication of the infection, emergence of resistant pathogens, or host immune deficiencies. This can lead to persistent inflammation, ongoing infection, or secondary complications such as subdural effusion or vasculitis, which contribute to prolonged or recurrent fever.

ELIGIBILITY:
Inclusion Criteria:

* Children from one month to 18 years.
* Who were diagnosed with bacterial meningitis or viral encephalitis and admitted to neurological department at Assiut University Children's Hospital (AUCH).
* Develop secondary or prolonged fever despite appropriate treatment.

Exclusion Criteria:

* Pediatric patients with suspected autoimmune encephalitis.
* Patient on immunosuppressive therapy (e.g., post-organ transplant, chemotherapy).
* Pediatric patients suspected metabolic disorders.
* Those with suspected endocrine dysfunction.

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Included children aged from one month to 18 years , who were diagnosed as bacterial meningitis or viral encephalitis and admitted to neurological department at AUCH and develop secondary or prolonged fever despite appropriate treatment .
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Causes of secondary and prolonged fever during treatment of bacterial meningitis and viral encephalitis | Basline
  Causes of secondary and prolonged fever during treatment of bacterial meningitis and viral encephalitis

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Mostafa Shafeek Khalaf Tawfeek, Professor of Pediatrics, Principal Investigator — Assiut University; Dr. Khalaf Abd El-Aal Sayed Mohamed, Lecturer of Pediatrics, Principal Investigator — Assiut University

REFERENCES:
- [Background] Brouwer MC, McIntyre P, de Gans J, Prasad K, van de Beek D. Corticosteroids for acute bacterial meningitis. Cochrane Database Syst Rev. 2010 Sep 8;(9):CD004405. doi: 10.1002/14651858.CD004405.pub3. PMID 20824838